CLINICAL TRIAL: NCT01648127
Title: Pharmacokinetics of Ceftaroline in Normal and Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Keith A. Rodvold (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Keith A. Rodvold, Professor, University of Illinois at Chicago
Organization: University of Illinois at Chicago (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TEF-MD-01
Record Dates: First submitted 2012-07-16; First posted 2012-07-24 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Drug Safety
Keywords: Ceftaroline; Pharmacokinetics; Obesity
MeSH Terms: conditions — Obesity | interventions — Ceftaroline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ceftaroline (Experimental): Ceftaroline intravenous 600 mg single dose
  Interventions: Drug: Ceftaroline

INTERVENTIONS:
Drug: Ceftaroline — A single dose of ceftaroline fosamil 600 mg as a 1-hour continuous intravenous infusion
  Other Names: Teflaro

SUMMARY:
The purpose of this study is to characterize plasma and urinary concentrations of ceftaroline following intravenous administration of a single dose of ceftaroline 600 mg in healthy subjects who are normal weight, overweight, and obese.

DETAILED DESCRIPTION:
This study is planned to be a Phase I, open-label, single period, single-dose pharmacokinetic study conducted in 32 healthy adult male and female subjects. Adult subjects will be recruited and assigned to one of four groups based on their body mass index and total body weight. Subject will receive a single dose of ceftaroline fosamil 600 mg as a 1-hour continuous intravenous infusion. Serial blood and urine samples will be collected over the next 12 hours to determine serum and urinary pharmacokinetics of ceftaroline. Safety evaluations will be assessed throughout the study and will include physical examination, vital sign monitoring, clinical laboratory tests (serum chemistry and hematology), pregnancy testing (female subjects only), monitoring of adverse events, and recording of concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult subjects
* nonsmokers within the last 1 year
* body mass index and total body weight within specific categories

Exclusion Criteria:

* history of significant hypersensitivity reaction or intolerance to ceftaroline or beta-lactam agents or heparin
* aspartate or alanine aminotransferase >3 times the upper limit of normal
* estimated creatinine clearance <60 mL/minute and serum creatinine >1.5 mg/dL
* female subjects who are pregnant or breast feeding
* history of alcohol or substance abuse or dependence within the last 1 year
* use of prescription or nonprescription drugs within last 7 to 14 days
* participations in a clinical trials within last 30 days
* donated blood (>500 mL) within the last 56 days

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of ceftaroline following intravenous administration of a single 600 mg dose to healthy subjects | 12 hours
  Plasma maximum serum concentration of ceftaroline Area-under-the-concentration-time curve of ceftaroline: Time frame Predose (time zero [0]) to 12 hours Total body clearance of ceftaroline Apparent volume of distribution of ceftaroline Elimination rate constant of ceftaroline Elimination half-life of ceftaroline Renal clearance of ceftaroline: Time frame Predose (time zero [0]) to 12 hours Amount of ceftaroline excreted in the urine: Time frame Predose (time zero [0]) to 12 hours

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of intravenous ceftaroline | 24 hours
  Number of participants with adverse events Number of participants with changes in clinical laboratories Number of participants with changes in vital sign assessments

CONTACTS AND LOCATIONS:
Overall Officials: Keith A Rodvold, Pharm.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Justo JA, Mayer SM, Pai MP, Soriano MM, Danziger LH, Novak RM, Rodvold KA. Pharmacokinetics of ceftaroline in normal body weight and obese (classes I, II, and III) healthy adult subjects. Antimicrob Agents Chemother. 2015 Jul;59(7):3956-65. doi: 10.1128/AAC.00498-15. Epub 2015 Apr 20. PMID 25896707